CLINICAL TRIAL: NCT03138278
Title: Impact on Family or Care-givers of Very Old ICU-survivors, Trajectories and 6 Months' Outcome in the Very Old.
Acronym: VIP2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer priority in the research group.
Sponsor: University of Bergen (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Principal Investigator, Hans Flaatten, Professor emeritus and senior consultant R&D, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ESICM VIP2
Record Dates: First submitted 2017-04-26; First posted 2017-05-03 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Functionally-Impaired Elderly; Caregivers; PTSD; Depression, Anxiety; Intensive Care Unit Syndrome
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Multicentre study with ≥ 100 ICUs from Europe. Randomisation at ICU level to give support to caregivers or not (cluster-randomisation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): ICU with ordinary care for elderly ICU survivors and their care-givers
- Telephone support (Active Comparator): ICU with day-time telephone support to care-givers
  Interventions: Other: Telephone support on demand

INTERVENTIONS:
Other: Telephone support on demand — Dedicated phone number for help and advice for caregivers
  Arms: Telephone support

SUMMARY:
It is known from extensive documentation that second victims in critical illness often are the care givers of the patients: family, friends or other persons. Although this has not been specifically studied in the very old patients, there is no reason to believe that this group will be different from other ICU patients. Even more so, in this very old age patient group there are seldom any older relatives. Partners, like wife/husband or other cohabitants, may be dead or themselves incapacitated. Many will be in institutional care. The closest care-givers will be middle-aged people such as children or others, if no partners are available.

The hypothesis is that critical illness can be a large stressor to care-givers of survivors in the VIP measured as the occurrence and severity of the usual problems like PTSD and depression. The investigators hypothesize that a low-threshold on-line support program decreases the magnitude of anxiety, depression and PTSD for care-givers of very old intensive care patients (VIP) after discharge.

DETAILED DESCRIPTION:
Aims of the study

* Results from family/care givers experience: Degree of involvement with post-ICU care, impact on their own health (depression, PTSD, burden questionnaire)
* Effect of a simple intervention: on-line support and/or telephone advice on Return to pre-ICU frailty score (patients) and Occurrence of PTSD and depression in care-givers
* Information on 6 months' outcome (frailty and mortality) in very old survivors after ICU in different European countries
* Information on trajectories in the time after discharge: Dead/alive, home, nursing home, new hospital admissions, living with family/other care-givers, etc.

ELIGIBILITY:
Inclusion Criteria:

* Hospital survivors after any ICU admission

Exclusion Criteria:

* Imminent terminal care

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Burden scale for Family Caregiver | 6 months post ICU discharge
  In order to assess the burden of care the investigaors will use an European questionaire developed within the EU and freely available online: Assessment of subjective burden of informal caregivers (http://www.psychiatrie.uk-erlangen.de/index.php?id=11049/) available in 20 European languages
Post traumatic stress (PTSD) in caregivers | 6 months post ICU discharge
  The study will use PTSD questionnaire PTSS-14 as described at www.sthk.nhs.uk/library/documents/7308450_ptss14.pdf.
Anxiety and Depression in caregivers | 6 months post ICU discharge
  The investigators will use the "Hospital anxiety and depression scale", a questionaire often used out of hospital as well. It is a simple questionaire that will be delivered to the care-givers after 6 months.

SECONDARY OUTCOMES:
6 months survival in the elderly ICU survivors | 6 months post ICU discharge
  Time of death in non-survivors (patients) will be sought through administrative hospital data (when available) or from care-givers
Trajectories in the elderly ICU survivors | 6 months post ICU discharge
  The investigators will seek to describe where the patients have been after hospital discharge: like rehabilitation facilities, nursing home, togehter with care-givers or in their own home.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Flaatten, Prof, Principal Investigator — University of bergen; ESICM

IPD SHARING:
Plan to Share IPD: No